CLINICAL TRIAL: NCT03809832
Title: Microbiologic Contamination of Home Non Invasive Ventilators
Acronym: MiCONIV
Status: Terminated | Type: Observational
Why Stopped: Preliminary results providing sufficient data
Sponsor: University Hospital, Rouen (Other)
Collaborators: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/363/OB
Record Dates: First submitted 2019-01-07; First posted 2019-01-18 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Respiratory Failure; COPD; Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients with COPD: Patients established on home non-invasive ventilation for COPD admitted for respiratory review will have a microbiological sampling of the ventilator humidifier
  Interventions: Diagnostic Test: Microbiological sampling
- Patients with OHS: Patients established on home non-invasive ventilation for obesity hypoventilation syndrome admitted for respiratory review will have a microbiological sampling of the ventilator humidifier
  Interventions: Diagnostic Test: Microbiological sampling

INTERVENTIONS:
Diagnostic Test: Microbiological sampling — An microbiological sampling of the ventilator humidifier will be performed.

SUMMARY:
Home non-invasive ventilators are daily used by patients with chronic respiratory failure. There are frequently used with warming and humidifying systems. These systems need to be cared for and frequently washed by the patient.

The aim of this study is to evaluate if the humidifying system of home ventilators are colonized by microbiological germs.

DETAILED DESCRIPTION:
The use of non-invasive ventilators is common for treating respiratory failure. Their care relies on the patients and their carers.

No study has assessed the efficacy of such care with respect to the number of microbiological specimens that remain in the humidifier.

ELIGIBILITY:
Inclusion Criteria:

* Patient established on home non invasive ventilation for more than 6 months
* With a compliance >4hours/day
* Who brought their ventilator for the assessment
* Diagnosed with COPD or Obesity hypoventilation syndrome (OHS)
* Who consent
* With an age > 18 years

Exclusion Criteria:

* Age under 18
* Ongoing exacerbation
* Not able to consent
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients established on long term home non-invasive ventilation admitted for a scheduled review.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of microbial contamination of non invasive ventilators humidifier | 7 days

SECONDARY OUTCOMES:
Microbiological ecology in the study population | 7 days
  The microbiological ecology of the ventilator humidifier will be describes (percentage of each pathogen)
Comparison between COPD and Obesity hypoventilation syndrome patients microbial ecology | 7 days
  We will compare the microbiological ecology of patients in the COPD and in the Obesity hypoventilation group (percentage of each pathogen in each group)
Compliance to recommendations regarding the maintenance of the humidifier | 7 days
  Compliance to recommendations will be assessed by a questionnaire containing 7 items regarding how the humidifier is maintained by the patient :
  * Who is maintaining the ventilator (descriptive)
  * At which frequency are you changing the water (Everyday (adequate), every other-day (almost adequate), every week (inadequate), more than weekly (inadequate)
  * What type of water are you using (descriptive)
  * At which frequency are you cleaning the mask (Everyday (adequate), every other-day (almost adequate), every week (inadequate), more than weekly (inadequate)
  * At which frequency are you cleaning the humidifier (Everyday (adequate), every other-day (almost adequate), every week (inadequate), more than weekly (inadequate)
  * How are you cleaning the humidifier? Water (inadequate), soap (adequate), dishawashing liquid (inadequate)
Correlation between compliance to maintenance recommendations and contamination rate | 7 days
Comparison of exacerbation frequency in COPD patients and isolation of respiratory pathogens in the humidifier | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Patout, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Bois-Guillaume, Normandy, France

IPD SHARING:
Plan to Share IPD: No